CLINICAL TRIAL: NCT00128115
Title: Proprietary Information - Exploratory (Non-Confirmatory) Trial
Brief Title: Treatment of Sarcopenia in Post-Hip Fracture Patients (0677-032)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0677-032; 2005_028
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — ibutamoren mesylate

INTERVENTIONS:
Drug: MK0677

SUMMARY:
The purpose of this study is to demonstrate an improvement in physical functional recovery, following administration of Drug for 24 weeks, in patients who have recently experienced a hip fracture. This study will also evaluate the safety and tolerability of Drug.

This is an early phase trial and some specific protocol information is proprietary and not publicly available at this time. (Full information is available to trial participants).

ELIGIBILITY:
Inclusion Criteria:

* Patient has had surgery for a unilateral hip fracture, and is considered to be partially or fully weight bearing after the surgery
* Surgical repair of the fracture has occurred no more than 4 days post hip fracture
* Prior to starting the study medication, the patient is enrolled in a rehabilitation program (as an in-patient or as an out-patient)
* Patient is judged to have been able to ambulate independently at home prior to their hip fracture (able to walk indoors in a familiar setting with little or no aid from another person)

Exclusion Criteria:

* Patient has an unstable medical condition
* Patient has a hip fracture that is due to bone pathology other than osteoporosis (e.g., malignancy, or Paget's Disease), or major trauma (e.g. motor vehicle accident).
* Patient has Type I diabetes
* Patient has Type II diabetes with any of conditions;

  1. Patient is currently taking more than one anti-hyperglycemic agent, or is taking a single combination anti-hyperglycemic drug containing more than one anti-hyperglycemic medication
  2. Patient is currently receiving insulin. Note: A short-term course of insulin required for glycemic control post hip fracture surgery is not exclusionary
  3. Patient has diabetic retinopathy
  4. Patient is unwilling or unable to monitor glucose at home
* Patient has been diagnosed with any neuromuscular or neurological disease causing muscle weakness
* Patient has cancer, or had a diagnosis of any malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or adequately treated in situ cervical cancer
* Patient has active carpal tunnel syndrome
* Patient was living in a nursing home prior to the hip fracture (Note: - Patients who were living in an assisted-living facility prior to the hip fracture are eligible for enrollment)
* Patient was permanently wheelchair bound prior to the hip fracture

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

SECONDARY OUTCOMES:
Proprietary Information - Exploratory (Non-Confirmatory) Trial

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- Msd Sharp & Dohme Gmbh, Haar, Germany
- MSD (Norge) AS, Drammen, Norway
- Merck Sharp & Dohme De Espana, S.A.E., Madrid, Madrid, Spain
- Merck Sharp & Dohme (Sweden) AB, Sollentuna, Sweden
- Merch Sharp & Dohme Ltd., Hoddesdon, Hertfordshire, United Kingdom

REFERENCES:
- [Derived] Adunsky A, Chandler J, Heyden N, Lutkiewicz J, Scott BB, Berd Y, Liu N, Papanicolaou DA. MK-0677 (ibutamoren mesylate) for the treatment of patients recovering from hip fracture: a multicenter, randomized, placebo-controlled phase IIb study. Arch Gerontol Geriatr. 2011 Sep-Oct;53(2):183-9. doi: 10.1016/j.archger.2010.10.004. Epub 2010 Nov 9. PMID 21067829